CLINICAL TRIAL: NCT00003914
Title: Phase II Study of Dolastatin-10 in Patients With Advanced Renal Cell Carcinoma
Brief Title: Dolastatin 10 in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry C. Pitot, M.D., Mayo Clinic
Purpose: Treatment
Other Study IDs: CDR0000067094; P30CA015083 (NIH); 975002 (Other: Mayo Clinic Cancer Center); T98-0024 (Other: NCI Protocol); 372-99 (Other: Mayo Clinic IRB)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — dolastatin 10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dolastatin 10

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dolastatin 10 in treating patients with advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate to dolastatin 10 in patients with advanced renal cell carcinoma. II. Describe the toxicities of this regimen in this patient population. III. Assess the development of peripheral neuropathy in this patient population using this regimen. IV. Assess a limited sampling of pharmacokinetics and correlate with toxicity in these patients.

OUTLINE: Patients receive dolastatin 10 IV every 3 weeks. Treatment continues for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients with documented complete response receive an additional 2 courses, and may receive retreatment at the time of progression at the discretion of the investigator. Patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study over 4-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed renal cell carcinoma considered incurable by surgery and not amenable to radiation therapy with curative intent Locally advanced disease OR Locally recurrent disease OR Metastatic disease No transitional cell carcinoma Measurable disease No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST less than 3 times upper limit of normal (ULN) Bilirubin normal Renal: Creatinine less than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease Metabolic: Oral intake at least 1,200 calories per day Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No uncontrolled infection No known seizure disorder No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No other medical or psychiatric condition that would interfere with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy No concurrent immunomodulating agents Chemotherapy: No prior chemotherapy for renal cell carcinoma No other concurrent cytostatic or cytotoxic therapy Endocrine therapy: At least 4 weeks since prior hormonal therapy No concurrent hormonal agents Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy No prior radiotherapy to greater than 15% of bone marrow No concurrent radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Pitot, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota